CLINICAL TRIAL: NCT01955681
Title: A Retrospective, Non-interventional Study to Evaluate EGFR-Tyrosine Kinase Inhibitor Retreatment in Patients With Locally Advanced or Metastatic EGFR Mutated NSCLC Who Previously Treated With EGFR-TKI as First-line Therapy and Chemotherapy as Second-line Therapy - SEQUENCE Study
Brief Title: A Retrospective, Non-interventional, Multicenter, Observational Chart Review Study to Explore the Clinical Benefits of Retreatment With TKI in the Real World.
Acronym: SEQUENCE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OTW-XXX-2013/1
Record Dates: First submitted 2013-09-30; First posted 2013-10-07 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Locally Advanced or Metastatic EGFR Mutated NSCLC.
Keywords: Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor retrement.

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective, non-interventional, multicenter, observational chart review study to explore the clinical benefits of retreatment with TKI in the real world.

DETAILED DESCRIPTION:
This study is designed to retrospectively review the medical and chemotherapy records of 300 patients with EGFR mutation positive adenocarcinoma NSCLC. Eligible patients are as follows: histologically or cytologically confirmed NSCLC, undergone EGFR-TKI retreatment sometime after the failure of the initial EGFR-TKI. After initial treatment, patients had been treated with chemotherapy and subsequently re-treated with EGFR-TKI will be identified. The target population will be derived from multicentre in Taiwan. The study aim is to evaluate clinical effect in re-administration of EGFR-TKI using retrospectively collected data from these eligible patients to provide valuable information.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with advanced adenocarcinoma or positive result of thyroid transcription factor 1 NSCLC
2. Positive Epidermal Growth Factor Receptor mutation result with sensitive mutation
3. Female or male aged ≧20 years
4. Patients treated with Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor and subsequently treated with chemotherapy before re-administration of Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor. Exclusion Criteria:

1. Patients with EGFR mutation status of positive exon 20 T790M mutation only. 2. Patients who are confirmed of squamous type NSCLC

Ages: 20 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic Epidermal Growth Factor Receptor mutated Non-small-cell Lung Cancer who Previously Treated with Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor as First-line therapy and chemotherapy as second-line Therapy - SEQUENCE study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The treatment duration of Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor re-administration | From the start of re-administration of EGFR-TKI to data cut-off date, assessed approximately up to 6 months.
  The median duration of re-administration of Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor will be summarized by days or months, if applicable. The range of this treatment duration will also be presented. All analyses will be performed on all eligible patients in this study.

SECONDARY OUTCOMES:
Assessment of progression-free survival for initial, second EGFR-TKI treatment and chemotherapy between two Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor treatments. | From the start of administration of EGFR-TKI to data cut-off date, assessed approximately up to 6 months.
  The outcome of progression-free survival will be presented with median values and associated 95% CIs by Kaplan-Meier curve. PFS is defined as the time interval (in weeks) from the start date of a given treatment to the date of disease progression or death, respectively, which one is observed first. Subjects who did not progress or die without a reported progression will be censored on the date of their last tumor assessment.
Assessment of overall survival for initial, second EGFR-TKI treatment and chemotherapy between two Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor treatments. | From the start of administration of EGFR-TKI to data cut-off date, assessed approximately up to 6 months.
  The outcome of overall survival will be presented with median values and associated 95% CIs by Kaplan-Meier curve. OS is defined as the time interval (in weeks) from the beginning of treatment until the date when death or lost to follow up is observed. For those subjects who have not died or lost to follow-up, survival duration will be censored at the last date the subject was known to be alive.
Assessment of response rate for initial, second EGFR-TKI treatment and chemotherapy between two Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor treatments. | From the start of administration of EGFR-TKI to data cut-off date, assessed approximately up to 6 months.
  The outcome about response rate and the proportion of response rate are estimated by all evaluable patients. The 95% exact confidence interval will be constructed around the rates. The best response during treatment sequences is determined in accordance with the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.
Assessment of disease control rate for initial, second EGFR-TKI treatment and chemotherapy between two Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor treatments. | From the start of administration of EGFR-TKI to data cut-off date, assessed approximately up to 6 months.
  The outcome of disease control rate are estimated by all evaluable patients. The 95% exact confidence interval will be constructed around the rates. Disease Control Rate is defined as patients who are respond to treatment (including CR-complete respond, PR-partial respond or SD- Stable Disease).
Record treatment duration in the initial EGFR-TKI therapy and first time chemotherapy. | Between the initial EGFR-TKI therapy and first time chemotherapy.
  Treatment duration in the initial EGFR-TKI therapy and first time chemotherapy.
Record the reason(s) for treatment change for initial and re-administration of EGFR-TKI therapy and first time chemotherapy (second-line treatment). | From the start of administration of EGFR-TKI to data cut-off date, assessed approximately up to 6 months.
  Record the reason(s) for treatment change for initial and re-administration of EGFR-TKI therapy and first time chemotherapy (second-line treatment).
Explore relationships between efficacy of EGFR-TKI initial and re-administration and patient characteristics or EGFR TKI treatment characteristics. | EGFR-TKI initial and re-administration
  Explore relationships between efficacy of EGFR-TKI initial and re-administration and patient characteristics (including demographics, histology, disease stage, sites of metastasis, ECOG PS) or EGFR TKI treatment characteristics (including EGFR mutation pattern, response to initial EGFR TKI or not, length of duration between first and second EGFR-TKI treatment)
overall survival (OS), plasma CEA level and chemotherapy regimens ever used. | between first time chemotherapy and EGFR-TKI re-administration
  Explore overall survival (OS), plasma CEA level and chemotherapy regimens ever used between first time chemotherapy and EGFR-TKI re-administration (including the types and number of chemotherapy regimens, and treatment duration) for those patients who have the above data available.
image peer review to evaluate tumour size retrospectively in different sequences of treatment | (1) initial and re-administration of EGFR-TKI therapy, (2) first time chemotherapy ever used (second-line treatment) after initial EGFR-TKI treatment.
  If the images are available, conduct image peer review to evaluate tumour size retrospectively in different sequences of treatment: (1) initial and re-administration of EGFR-TKI therapy, (2) first time chemotherapy ever used (second-line treatment) after initial EGFR-TKI treatment. Peer review time point includes baseline, best response and progression of last image while stopping treatment at each treatment mentioned above.
The reason(s) for the treatment change for initial and re-administration of EGFR-TKI therapy and first time chemotherapy (second-line treatment) after peer review | Initial and re-administration of EGFR-TKI therapy and first time chemotherapy (second-line treatment) after peer review.
  Evaluate the reason(s) for the treatment change for initial and re-administration of EGFR-TKI therapy and first time chemotherapy (second-line treatment) after peer review and compare the difference of reason(s) for the treatment change between initiatial evaluation and after peer review.

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Min Chen, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Gee-Chen Chang, Principal Investigator — Veterans General Hospital -Taichung; Chong-Jen Yu, Principal Investigator — National Taiwan University Hospital; Cheng-Ta Yang, Principal Investigator — Chang Gung Memorial Hospital; Te-Chun Hsia, Principal Investigator — China Medical University Hospital; Meng-Chih Lin, Principal Investigator — Chang-Gung Memorial Hospital Kaohsiung; Ying-Huang Tsai, Principal Investigator — Chang Gung Memorial Hospital, Chiayi
Locations (6):
- Taiwan (6):
  - Chiayi City
  - Kaohsiung City
  - Taichung
  - Research Site, Taipei
  - Taipei
  - Taoyuan District

REFERENCES:
- See also: CSR_Synopsis_NIS-OTW-XXX-2013_1 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1850&filename=CSR_NIS-OTW-XXX-2013_1.pdf